CLINICAL TRIAL: NCT06976099
Title: Multicenter Prospective Cohort Study of Hypertriglyceridemia Acute Pancreatitis
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, wen li, MD, Director, Biomarker Discovery and Validation Platform, Translational Medicine National Major Science and Technology Infrastructure at PUMCH, Peking Union Medical College Hospital
Other Study IDs: K5714
Record Dates: First submitted 2025-03-10; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Acute Pancreatitis (AP); Hypertriglyceridemia Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood: 1 purple-topped tube x 4mL (EDTA anticoagulant plasma separation tube) and 1 red-topped/yellow-topped tube x 4mL (serum separation tube) Fresh Urine: 10 mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Hypertriglyceridemia-associated acute pancreatitis (HTG-AP) is the second leading cause in China and is receiving increasing global attention. Research on HTG-AP has been hindered by the heterogeneity and complexity of the disease, as well as the limitations of prior single-center studies with small sample sizes, inadequate collection of clinical data, lack of sustainable follow-up, and insufficient tools for large-scale data collection, analysis, and biomarker testing. To address these unique challenges and leverage the opportunity to gain a deeper understanding of HTG-AP, the China Hypertriglyceridemia Pancreatitis Study Group (CHPSG) was initiated in April 2023 as a multi-center collaboration. By utilizing the advantages of multi-center studies, such as external validity and larger sample sizes, CHPSG aims to investigate the prevalence, clinical characteristics, natural history, and risk factors of HTG-AP in China. The consortium will also explore the differences between HTG-AP and other etiologies of pancreatitis, with an emphasis on systemic and local complications, recurrence, and long-term quality of life. Through its phased approach, CHPSG seeks to develop targeted strategies for the prevention and treatment of HTG-AP, ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years;
* Diagnosed with AP based on at least two of the following criteria (1) acute onset of upper abdominal pain; (2) more than three times the upper limit of the normal range of serum lipase or amylase levels; and (3) typical radiological findings of AP on computed tomography (CT), magnetic resonance imaging, or ultrasonography;
* HTG with serum triglyceride levels >500 mg/dL (5.65 mmol/L) during the current AP episode or at admission;
* Patients must have good compliance, with the ability and willingness to adhere to study protocols, provide written informed consent, and maintain their current lifestyle during the study period

Exclusion Criteria:

* History of chronic pancreatitis or pancreatic cancer;
* Severe comorbidities such as malignancy, acute myocardial infarction, or extensive cerebral infarction;
* Prior use of lipid-lowering medications;
* Pregnancy or breastfeeding;
* Lack of signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with AP based on at least two of the following criteria (1) acute onset of upper abdominal pain; (2) more than three times the upper limit of the normal range of serum lipase or amylase levels; and (3) typical radiological findings of AP on computed tomography (CT), magnetic resonance imaging, or ultrasonography
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of organ dysfunction | 1-2 weeks
  Assessment of multi-organ dysfunction syndrome (MODS), acute respiratory distress syndrome (ARDS), acute kidney injury (AKI), and other complications
Clinical outcomes | 1-2 weeks
  Hospital length of stay, ICU admission rate, and mortality
Incidence of recurrent HTG-AP | 1 year
  The recurrence rate within a defined period
Risk factors for recurrence | 1 year
  Identification of factors such as triglyceride (TG) levels, BMI, diabetes status, medication use, and lifestyle habits.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share individual participant data due to privacy regulations and ethical considerations.